CLINICAL TRIAL: NCT01715337
Title: Effects of Pulmonary Rehabilitation on Muscle Fibre Composition and Capillaries in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Effects of Rehabilitation on Muscle Fibre Composition and Capillaries in Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Collaborators: German Sport University, Cologne (Other)
Responsible Party: Principal Investigator, Klaus Kenn, Head physician (department of pneumology), Schön Klinik Berchtesgadener Land
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: COPD muscle 2011
Record Dates: First submitted 2012-10-24; First posted 2012-10-26 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: muscle fibre; capillary; rehabilitation; exercise training
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pulmonary rehabilitation (Other)
  Interventions: Other: pulmonary rehabilitation

INTERVENTIONS:
Other: pulmonary rehabilitation — 3-week rehabilitation including exercise training, breathing therapy, psychosocial support, medical treatment etc.

SUMMARY:
Pulmonary rehabilitation has been established as an evidence-based and recommended therapy in patients with chronic obstructive pulmonary disease (COPD). The aim of our study is to show a potential change in muscle fibre composition and in the amount of capillaries in quadriceps muscle from pre tob post 3-week rehabilitation. Pulmonary rehabilitation includes standardised exercise training, e.g. cycling and strength training for major muscle groups.

ELIGIBILITY:
Inclusion Criteria:

* chronic obstructive pulmonary disease
* FEV1%pred. < 50%

Exclusion Criteria:

* acute exacerbation
* exacerbation in the last 4 weeks

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-02; Primary Completion 2013-03 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Change in the amount of capillaries in muscle fibre type I | change from pre (day 1) to post rehabilitation (day 21)

SECONDARY OUTCOMES:
Change in the amount of capillaries in muscle fibre type IIa | Change from pre (day 1) to post rehabilitation (day 21)
Change in the cross-sectional area of muscle fibre type I | Change from pre (day 1) to post rehabilitation (day 21)
Change in the cross-sectional area of muscle fibre type IIa | Change from pre (day 1) to post rehabilitation (day 21)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Kenn, Dr. med., Study Chair — Klinikum Berchtesgadener Land
Locations (1):
- Schön Klinik Berchtesgadener Land, Schönau am Königssee, Germany